CLINICAL TRIAL: NCT05495477
Title: Effects of Non-invasive Ventilation (NIV) and Continuous Positive Airway Pressure (CPAP) on Ventilation Distribution, Measured by Electrical Impedance Tomography (EIT), During Deep Sedation in Paediatric Patients
Brief Title: Effects of NIV and CPAP on Ventilation Distribution, Measured by EIT, During Deep Sedation in Paediatric Patients
Acronym: NIVEIT-ped
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/2178
Record Dates: First submitted 2022-02-25; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Failure; Sedation; Mechanical Ventilation Complication
Keywords: NIV; CPAP; EIT;
MeSH Terms: conditions — Respiratory Insufficiency; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spontaneous breathing (Active Comparator): Electrical impedance tomography (EIT).
  Interventions: Device: EIT
- CPAP mode (Active Comparator): Electrical impedance tomography (EIT).
  Interventions: Device: EIT
- NIV- S/T mode (Active Comparator): Electrical impedance tomography (EIT).
  Interventions: Device: EIT

INTERVENTIONS:
Device: EIT — Evaluation of ventilation distrinution during deep sedation through EIT

SUMMARY:
In patients undergoing spontaneous breathing (SB) deep sedation there is a re-distribution of ventilation towards lungs non-dependant areas (ventral areas in supine position).

Non-invasive ventilation (NIV), offering positive pressure, should favour a better ventilation of dependant areas (dorsal areas in supine position), making ventilation more homogeneous and increasing functional residual capacity.

Electrical impedance tomography (EIT) is a non-invasive, non-operator dependent, bedside, radiations-free diagnostic tool, feasible in paediatric patients and repeatable; it allows to study ventilation distribution, and it can measure and calculate also parameters that are related to the homogeneity of ventilation and the response to certain therapeutic maneuvers, such as anaesthesia or PEEP-application.

Uses of EIT in paediatric age are described in literature, but it has never been described as being used in Non-Operating Room Anaesthesia, nor in other cases of SB deep sedation. In addition, the impact of NIV on the distribution of ventilation in healthy paediatric patients undergoing deep sedation has never been described.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric age (from 1 to 10 years old)
* ASA score ≤ 2
* Sedation time ≥ 30 min

Exclusion Criteria:

* ASA score ≥ 3
* Lung pathologies (such as asthma, bronchopulmonary dysplasia, obstructive sleep apnoea) Preterm infant
* Severe obesity
* Dorso-lumbar pathologies or other bone pathologies associated with restrictive lung disease (such as scoliosis, kyphosis)
* Neuromuscular, mitochondrial, metabolic or chromosomal disease with hypotonia
* CPAP or NIV treatment at home
* Hand-Bag Ventilation (HBV) during the procedure (loss of the respiratory drive)
* Non-Total IntraVenous Anaesthesia (TIVA), adherence to the sedation protocol
* Implantable devices not compatible with EIT (such as pace-makers and implantable cardioverter defibrillator)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-06-28 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Regional Ventilation Delay (pixels %), RDV | 1 day
  It's an index of atelectrauma, supra-distension and in general an inhomogeneous ventilation

SECONDARY OUTCOMES:
Inhomogeneity Index (pixels), GI | 1 day
Gravity Centre(pixels %), GC | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Chidini, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leonhardt S, Lachmann B. Electrical impedance tomography: the holy grail of ventilation and perfusion monitoring? Intensive Care Med. 2012 Dec;38(12):1917-29. doi: 10.1007/s00134-012-2684-z. Epub 2012 Sep 20. PMID 22992946
- [Background] Zhao Z, Moller K, Steinmann D, Frerichs I, Guttmann J. Evaluation of an electrical impedance tomography-based Global Inhomogeneity Index for pulmonary ventilation distribution. Intensive Care Med. 2009 Nov;35(11):1900-6. doi: 10.1007/s00134-009-1589-y. Epub 2009 Aug 4. PMID 19652949
- [Background] Spinelli E, Mauri T, Fogagnolo A, Scaramuzzo G, Rundo A, Grieco DL, Grasselli G, Volta CA, Spadaro S. Electrical impedance tomography in perioperative medicine: careful respiratory monitoring for tailored interventions. BMC Anesthesiol. 2019 Aug 7;19(1):140. doi: 10.1186/s12871-019-0814-7. PMID 31390977
- [Background] Bordes J, Goutorbe P, Cungi PJ, Boghossian MC, Kaiser E. Noninvasive ventilation during spontaneous breathing anesthesia: an observational study using electrical impedance tomography. J Clin Anesth. 2016 Nov;34:420-6. doi: 10.1016/j.jclinane.2016.04.016. Epub 2016 Jun 16. PMID 27687426
- [Background] Humphreys S, Pham TM, Stocker C, Schibler A. The effect of induction of anesthesia and intubation on end-expiratory lung level and regional ventilation distribution in cardiac children. Paediatr Anaesth. 2011 Aug;21(8):887-93. doi: 10.1111/j.1460-9592.2011.03547.x. Epub 2011 Mar 14. PMID 21395895
- [Derived] Chidini G, Marchesi T, Catenacci SS, Florio G, Conti G, Lanni S, Filocamo G, Patria F, Guerrini M, Milani G, Grasselli G. Effects of Noninvasive Respiratory Support on Ventilation Distribution During Spontaneous Breathing Sedation in Preschool/School-Aged Children: An Electrical Impedance Tomography Study. Paediatr Anaesth. 2025 Jul;35(7):562-572. doi: 10.1111/pan.15098. Epub 2025 Mar 22. PMID 40119601